CLINICAL TRIAL: NCT00169143
Title: Study of R-ACVBP Regimen Supported by Pegfilgrastim in Previously Untreated Patients Aged From 18 to 60 Years With High-Risk Diffuse Large B-Cell Lymphoma (Age-adjusted Ipi >or= 2)
Brief Title: Study of R-ACVBP Regimen Supported by Pegfilgrastim in High-Risk Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Collaborators: Amgen (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNH 03-39B
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Untreated CD20-positive Large B-cell Lymphoma
Keywords: Diffuse large B cell lymphoma; Pegfilgrastim; Autotransplant
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; LNH 87 protocol; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rituximab + ACVBP regimen plus Pegfilgrastim
Procedure: Autologous stem cell transplant

SUMMARY:
Evaluation of the efficacy of a single injection of Pegfilgrastim (6mg) administered at day 3 of each cycle of R-ACVBP regimen during 4 cycles in patients with CD20+ diffuse large B-cell lymphoma presenting at least 2 adverse prognostic factor of the age-adjusted international prognostic index (Aa-IPI).

DETAILED DESCRIPTION:
This is a phase II, multicentric, open-label, non-randomized study, evaluating the efficacy of a single injection of Pegfilgrastim (6mg) administered at day 3 of each cycle of R-ACVBP regimen during 4 cycles in patients aged 18 to 60 years with previously untreated CD20+ diffuse large B-cell lymphoma presenting at least 2 adverse prognostic factor of the age-adjusted international prognostic index (Aa-IPI), and eligible for transplant.

It is anticipated that 60 subjects will be enrolled over 2 years (from 2004 to 2006), in a group sequential manner one planned interim analysis.

The duration of the treatment period is approximately 26 weeks and patients are followed until Death.

The total Duration of the study is expected to be 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically proven CD20+ diffuse large B cell lymphoma (WHO Classification).
* Age >18 and < 61 years, eligible for transplant.
* Patient not previously treated.
* With at least two prognostic factors of the Aa-IPI.
* With a minimum life expectancy of 3 months.
* Creatinin level ≤ 150mmol/l, total bilirubin level 30mmol/l and transaminases 2.5 maximum normal level, unless abnormalities are related to the lymphoma.
* Neutrophils > 1.5 G/l and platelets > 100 G/l, unless if patient has a bone marrow infiltration.
* Negative HIV, HBV and HCV serologies 4 weeks (except after vaccination).
* Having previously signed a written informed consent.

Exclusion Criteria:

* Any other histological type of lymphoma.
* Any history of treated or non-treated indolent lymphoma.
* Central nervous system or meningeal involvement by lymphoma.
* Contra-indication to any drug contained in the chemotherapy regimens.
* Any history of cancer during the last 5 years, with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma.
* Any serious active disease (according to the investigator's decision).
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study.
* Pregnant or lactating women or women of childbearing potential not currently practicing an adequate method of contraception.
* Adult patient under tutelage.

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60
Dates: Start 2004-05 (Actual); Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the optimal combined dose intensity of the drug regimen

SECONDARY OUTCOMES:
Specific dose intensities, incidence of neutropenia and neutropenic fever, duration of severe neutropenia, complete response rate, event-free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Haioun, MD, Study Chair — Hôpital Henri Mondor, Créteil, France
Locations (6):
- France (6):
  - Hôpital Henri Mondor, Créteil
  - Service d'Hématologie Clinique - CHU Le Bocage, Dijon
  - Hôpital Saint Louis, Paris
  - Service d'Hématologie - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - CHRU de Nancy Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Green MD, Koelbl H, Baselga J, Galid A, Guillem V, Gascon P, Siena S, Lalisang RI, Samonigg H, Clemens MR, Zani V, Liang BC, Renwick J, Piccart MJ; International Pegfilgrastim 749 Study Group. A randomized double-blind multicenter phase III study of fixed-dose single-administration pegfilgrastim versus daily filgrastim in patients receiving myelosuppressive chemotherapy. Ann Oncol. 2003 Jan;14(1):29-35. doi: 10.1093/annonc/mdg019. PMID 12488289
- [Background] Holmes FA, O'Shaughnessy JA, Vukelja S, Jones SE, Shogan J, Savin M, Glaspy J, Moore M, Meza L, Wiznitzer I, Neumann TA, Hill LR, Liang BC. Blinded, randomized, multicenter study to evaluate single administration pegfilgrastim once per cycle versus daily filgrastim as an adjunct to chemotherapy in patients with high-risk stage II or stage III/IV breast cancer. J Clin Oncol. 2002 Feb 1;20(3):727-31. doi: 10.1200/JCO.2002.20.3.727. PMID 11821454
- [Background] Vose JM, Crump M, Lazarus H, Emmanouilides C, Schenkein D, Moore J, Frankel S, Flinn I, Lovelace W, Hackett J, Liang BC. Randomized, multicenter, open-label study of pegfilgrastim compared with daily filgrastim after chemotherapy for lymphoma. J Clin Oncol. 2003 Feb 1;21(3):514-9. doi: 10.1200/JCO.2003.03.040. PMID 12560443
- [Background] Haioun C, Lepage E, Gisselbrecht C, Salles G, Coiffier B, Brice P, Bosly A, Morel P, Nouvel C, Tilly H, Lederlin P, Sebban C, Briere J, Gaulard P, Reyes F. Survival benefit of high-dose therapy in poor-risk aggressive non-Hodgkin's lymphoma: final analysis of the prospective LNH87-2 protocol--a groupe d'Etude des lymphomes de l'Adulte study. J Clin Oncol. 2000 Aug;18(16):3025-30. doi: 10.1200/JCO.2000.18.16.3025. PMID 10944137
- [Derived] Copie-Bergman C, Cuilliere-Dartigues P, Baia M, Briere J, Delarue R, Canioni D, Salles G, Parrens M, Belhadj K, Fabiani B, Recher C, Petrella T, Ketterer N, Peyrade F, Haioun C, Nagel I, Siebert R, Jardin F, Leroy K, Jais JP, Tilly H, Molina TJ, Gaulard P. MYC-IG rearrangements are negative predictors of survival in DLBCL patients treated with immunochemotherapy: a GELA/LYSA study. Blood. 2015 Nov 26;126(22):2466-74. doi: 10.1182/blood-2015-05-647602. Epub 2015 Sep 15. PMID 26373676
- See also: Official site of the Groupe d'Etude des Lymphomes de l'Adulte (In french) — http://www.gela.org